CLINICAL TRIAL: NCT01518309
Title: An Open-Label Safety Study of Pimavanserin in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACP-103-010
Record Dates: First submitted 2008-12-16; First posted 2012-01-26 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pimavanserin tartrate (ACP-103) (Experimental): Tablets taken once daily by mouth at 20, 40, or 60 mg doses
  Interventions: Drug: pimavanserin tartrate (ACP-103)

INTERVENTIONS:
Drug: pimavanserin tartrate (ACP-103) — Tablets taken once daily by mouth at 20, 40, or 60 mg doses

SUMMARY:
This is an open-label extension study to assess the long-term safety and tolerability of pimavanserin (ACP-103) in subjects with Parkinson's Disease Psychosis (PDP).

ELIGIBILITY:
Inclusion Criteria-

* Patients of any age, male or female with a clinical diagnosis of idiopathic Parkinson's disease, who participated in a previous (Phase II) clinical trial that evaluated pimavanserin
* Patients who may, in the opinion of the treating physician, benefit from continued therapy with pimavanserin
* Patient is willing and able to provide consent

Exclusion Criteria-

* Female patient of childbearing potential
* Patient has a clinically significant concurrent medical illness
* Patient is judged by the treating physician to be inappropriate for the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-11-17 (Actual); Primary Completion 2013-05-02 (Actual); Study Completion 2013-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Danbury, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension study, including patients with idiopathic Parkinson's Disease (PD) who had completed study ACP-103-006 (PD psychosis [PDP]) or study ACP-103-004 (PD with dyskinesias) and would benefit from continued pimavanserin treatment, as judged by the investigator.
Groups:
- Pimavanserin: All patients started treatment with pimavanserin 20 mg/day. Based on clinical benefit and Investigator judgment, dose escalation to 40 mg and 60 mg was allowed, after a minimum of 2 and 4 weeks treatment duration, respectively. Dose reductions to 40 and/or 20 mg/day were allowed for the management of AEs or intolerability.
Period: Overall Study
Arm/Group | Pimavanserin
Started | 39
Completed | 0
Not Completed | 39
Not completed — Adverse Event | 6
Not completed — Death | 6
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 3
Not completed — Sponsor Decision | 2
Not completed — Not in Predefined Categories | 9

BASELINE CHARACTERISTICS:
Arm/Group | Pimavanserin
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 38
  Hispanic/Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 39
Clinical Global Impression of Severity [Mean (Standard Deviation); unit: Score on a scale] — The Clinical Global Impression-Severity (CGI-S) Scale is a 1-item scale, used to rate the severity of the disorder from 0 (not assessed) to 7 (among the most extremely ill patients). A higher CGI-S score denotes more severe depression.
  Score on a scale | 3.6 (0.22)
UPDRS tremor [Median (Full Range); unit: Score on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) tremor score range was 0 (absent) to 4 (marked; interferes with most activities).
  Score on a scale | 1.0 [0 to 3]
UPDRS duration of dyskinesias [Median (Full Range); unit: Score on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) duration of dyskinesias score was 0 (none) to 4 (76-100% present during the waking day).
  Score on a scale | 0.0 [0 to 3]
UPDRS disability of dyskinesias [Median (Full Range); unit: Score on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) disability of dyskinesias score was 0 (not disabling) to 4 (completely disabling).
  Score on a scale | 0.0 [0 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Patients With Drug-related Treatment-emergent Adverse Events (AEs)
Description: Number (%) of patients with drug-related treatment-emergent AEs
Time Frame: From first to last study drug dose plus 30 days
Population: Patients treated with at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin
Number analyzed (Participants) | 39
Participants | 17

ADVERSE EVENTS:
Time Frame: Study treatment (median treatment duration: 475 days)
Arm/Group | Pimavanserin
All-Cause Mortality (participants affected / at risk) | 8/39
Serious Adverse Events (participants affected / at risk) | 18/39
Other Adverse Events (participants affected / at risk) | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=39)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2)
Hip fracture (Injury, poisoning and procedural complications) | 3 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=39)
Anaemia (Blood and lymphatic system disorders) | 8 (10)
Constipation (Gastrointestinal disorders) | 9 (13)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 3 (4)
Asthenia (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 5 (7)
Pain (General disorders) | 3 (3)
Cellulitis (Infections and infestations) | 3 (4)
Urinary tract infection (Infections and infestations) | 8 (14)
Contusion (Injury, poisoning and procedural complications) | 4 (7)
Fall (Injury, poisoning and procedural complications) | 7 (12)
Skin laceration (Injury, poisoning and procedural complications) | 3 (5)
Prothrombin time prolonged (Investigations) | 5 (5)
Weight decreased (Investigations) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6)
Groin pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Confusional state (Nervous system disorders) | 6 (6)
Dyskinesia (Nervous system disorders) | 4 (4)
Somnolence (Nervous system disorders) | 5 (7)
Agitation (Psychiatric disorders) | 4 (5)
Depression (Psychiatric disorders) | 5 (6)
Hallucination (Psychiatric disorders) | 9 (10)
Hallucination, visual (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)
Orthostatic hypertension (Vascular disorders) | 5 (9)
Faecaloma (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 2 (3)
Blood bilirubin increased (Investigations) | 2 (3)
Haematocrit decreased (Investigations) | 2 (2)
Haemoglobin decreased (Investigations) | 2 (2)
Low density lipoprotein increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (4)
Pyuria (Investigations) | 2 (2)
Retyculocyte count decreased (Investigations) | 2 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Facial wasting (Metabolism and nutrition disorders) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Amnesia (Nervous system disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2)
Dementia (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (4)
Dystonia (Nervous system disorders) | 2 (3)
Gait disturbance (Nervous system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Delusion (Psychiatric disorders) | 2 (2)
Paranoia (Psychiatric disorders) | 2 (2)
Sleep disorder (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 2 (2)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.